CLINICAL TRIAL: NCT05997368
Title: Investigation of the Relationship of Pain Perception and Pain Belief With Age in People With Chronic Lack Pain
Status: Completed | Type: Observational
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, assistant professor, Uskudar University
Other Study IDs: Uskudar67
Record Dates: First submitted 2023-08-09; First posted 2023-08-18 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Chronic Pain; Low Back Pain
Keywords: pain perception; pain beliefs
MeSH Terms: conditions — Chronic Pain; Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- young group: Participants aged 18-39
  Interventions: Other: Survey1
- middle-aged group: Participants aged 40-56
  Interventions: Other: Survey2
- elderly group: Participants aged 57-79
  Interventions: Other: Survey3

INTERVENTIONS:
Other: Survey1 — As a research, it was planned to be a quantitative research. Data collection will be conducted through online and face-to-face surveys. Scales and forms to be found and used in the research: The Pain Beliefs Questionnaire-PBQ, Numerical Rating Scale (NRS-11) and The Central Of Pain Scale-COPS. By handing out the paper format to the participants and uploading it to the Google Forms system online, it can be downloaded from mail, social media or mobile phone applications such as message, Mail, etc. They will be asked to participate in the study by accessing
  Groups: young group
Other: Survey2 — As a research, it was planned to be a quantitative research. Data collection will be conducted through online and face-to-face surveys. Scales and forms to be found and used in the research: The Pain Beliefs Questionnaire-PBQ, Numerical Rating Scale (NRS-11) and The Central Of Pain Scale-COPS. By handing out the paper format to the participants and uploading it to the Google Forms system online, it can be downloaded from mail, social media or mobile phone applications such as message, Mail, etc. They will be asked to participate in the study by accessing
  Groups: middle-aged group
Other: Survey3 — As a research, it was planned to be a quantitative research. Data collection will be conducted through online and face-to-face surveys. Scales and forms to be found and used in the research: The Pain Beliefs Questionnaire-PBQ, Numerical Rating Scale (NRS-11) and The Central Of Pain Scale-COPS. By handing out the paper format to the participants and uploading it to the Google Forms system online, it can be downloaded from mail, social media or mobile phone applications such as message, Mail, etc. They will be asked to participate in the study by accessing
  Groups: elderly group

SUMMARY:
This study was planned to investigate the relationship between pain perceptions and pain beliefs of individuals in different age groups with chronic low back pain and symptom severity.

DETAILED DESCRIPTION:
The study will be conducted as an observational descriptive and cross-sectional research. Participants will be recruited after the purpose and content of the research are explained by the researchers, their written consent is read, and the volunteers who agree to be included in the study are given their written consent. The data collection process was carried out face-to-face and via a Google Forms survey over the internet, and will be conducted with the participants face-to-face and online. In the study; The pain beliefs questionnaire (PBQ), the centrality of pain scale (COPS) and the numerical rating scale (NRS-11) will be used.

ELIGIBILITY:
Inclusion Criteria:

* having low back pain for at least the past three months
* be between the ages of 18-79.

Exclusion Criteria:

* Those outside the age limit of 18-79 and illiteracy.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will take place in Istanbul, Turkey. Volunteers who accepted the voluntary consent form will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-09-02 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
The numeric rating scale - NRS-11 | 2 weeks
  When using the NRS-11, patients are asked to rate their pain on a scale of 0 to 10; where using integers (11 integers including zero) 0 represents "no pain" and 10 represents "worst possible pain". Based on prior studies and clinical experience of use, pain screening scores NRS-11 scores as mild (1-3) are classified as moderate (4-6) or severe (7-10).
The centrality of pain scale - COPS) | 2 weeks
  It is a short 10-item self-report scale designed to assess the centrality of pain. COPS scores are significantly correlated with the clinician's assessment of individual-reported pain severity, disability, mental health, quality of life, and how well the patient's pain is controlled. Each item is rated on a five-point Likert scale. It is a 10-item questionnaire (1: strongly disagree, 2: disagree, 3: neither agree nor disagree, 4: agree, 5: strongly agree). Items 2, 4 and 9 are evaluated in reverse. The resulting value is the sum of all item scores. Higher scores indicate more "central" pain. The highest possible score is 50 and the lowest possible score is 10.
The pain beliefs questionnaire - PBQ | 2 weeks
  Two subtests of the test were created: the 8-item Organic Beliefs subtest and the 4-item Psychological Beliefs subtest. The item numbers of both subtests are listed as follows:
  Organic Beliefs: items 1, 2, 3, 5, 7, 8, 10, 11, Psychological Beliefs: Items 4, 6, 9, 12. The test takers are asked to indicate the most appropriate one for the participants from 6 options ranging from 1st "never" to 6th "always". The marked scores range from 1 to 6 for each item. The score collected for each subtest is calculated by taking the items in that subtest and summing them up and dividing the numbers by the number of items related to that subtest. An increase in the value calculated from the sub-dimension of the scale indicates that the belief in pain belonging to the sub-dimension is high, and a decrease in the value indicates low pain belief in the sub-dimension.

CONTACTS AND LOCATIONS:
Overall Officials: Mahsun EKİNCİ, Study Chair — Uskudar University
Locations (1):
- Üsküdar Unıversıty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] La Touche R, Grande-Alonso M, Arnes-Prieto P, Paris-Alemany A. How Does Self-Efficacy Influence Pain Perception, Postural Stability and Range of Motion in Individuals with Chronic Low Back Pain? Pain Physician. 2019 Jan;22(1):E1-E13. PMID 30700075
- [Background] Baird AJ, Haslam RA. Exploring differences in pain beliefs within and between a large nonclinical (workplace) population and a clinical (chronic low back pain) population using the pain beliefs questionnaire. Phys Ther. 2013 Dec;93(12):1615-24. doi: 10.2522/ptj.20120429. Epub 2013 Jul 25. PMID 23886843
- [Background] Pulvers K, Hood A. The role of positive traits and pain catastrophizing in pain perception. Curr Pain Headache Rep. 2013 May;17(5):330. doi: 10.1007/s11916-013-0330-2. PMID 23512722
- [Background] Walsh DA, Radcliffe JC. Pain beliefs and perceived physical disability of patients with chronic low back pain. Pain. 2002 May;97(1-2):23-31. doi: 10.1016/s0304-3959(01)00426-2. PMID 12031776
- [Background] Wandner LD, Scipio CD, Hirsh AT, Torres CA, Robinson ME. The perception of pain in others: how gender, race, and age influence pain expectations. J Pain. 2012 Mar;13(3):220-7. doi: 10.1016/j.jpain.2011.10.014. Epub 2012 Jan 5. PMID 22225969